CLINICAL TRIAL: NCT00850239
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate Safety and Efficacy of Dutogliptin/PHX1149T in Subjects With Type 2 Diabetes Mellitus on a Background Medication of Metformin
Brief Title: Safety and Efficacy Study of Dutogliptin/PHX1149T in Subjects With Type 2 Diabetes Mellitus on a Background Medication of Metformin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Phenomix (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Hans-Peter Guler, MD, Phenomix Corporation
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: PHX1149-PROT302
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; DPP4 inhibitor; dutogliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dutogliptin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): dutogliptin/PHX1149T
  Interventions: Drug: dutogliptin
- 2 (Placebo Comparator): Plabeco
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: dutogliptin — 400 mg
  Other Names: PHX1149T
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the efficacy of dutogliptin over 26 weeks (as evidenced by placebo-corrected changes in HbA1c relative to baseline), to demonstrate safety and tolerability of dutogliptin, and to demonstrate changes in fasting plasma glucose over 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed at least 4 months prior to Screening (Visit 1)
* Age 18 to 85 years, inclusive.
* Male and non-pregnant, non-lactating (and not planning to become pregnant during the study) female subjects with a BMI of 20 to 48 kg/m2, inclusive
* Current treatment of Type 2 diabetes mellitus with a stable dose of metformin of ≥ 2000 mg (or the highest tolerated dose) used in accordance with product labeling for at least 6 weeks prior to screening (Visit 1)
* HbA1c 7.0% - 10.0%, inclusive; and fasting plasma C peptide greater than 0.26 nmol/L (> 0.8 ng/mL; > 281 pmol/L) at screening (Visit 1)

Exclusion Criteria:

* Type 1 diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Primary objective is to demonstrate the efficacy of dutogliptin, as evidenced by placebo-corrected changes in HbA1c relative to baseline. | 26 weeks

SECONDARY OUTCOMES:
Demonstrate safety and tolerability of dutogliptin | 26 weeks
• Demonstrate changes in fasting plasma glucose | 26 weeks

CONTACTS AND LOCATIONS:
Locations (97):
- United States (34):
  - Phenomix Investigational Site 115, Montgomery, Alabama
  - Phenomix Investigational Site 121, Tempe, Arizona
  - Phenomix Investigational Site 137, Tempe, Arizona
  - Phenomix Investigational Site 105, Anaheim, California
  - Phenomix Investigational Site 123, Chico, California
  - Phenomix Investigational Site 134, Escondido, California
  - Phenomix Investigational Site 103, Long Beach, California
  - Phenomix Investigational Site 106, Los Angeles, California
  - Phenomix Investigational Site 143, Coral Gables, Florida
  - Phenomix Investigational Site 142, Hialeah, Florida
  - Phenomix Investigational Site 119, Jacksonville, Florida
  - Phenomix Investigational Site 133, Kissimmee, Florida
  - Phenomix Investigational Site 141, Dunwoody, Georgia
  - Phenomix Investigational Site 101, Honolulu, Hawaii
  - Phenomix Investigational Site 135, Chicago, Illinois
  - Phenomix Investigational Site 124, Indianapolis, Indiana
  - Phenomix Investigational Site 127, Indianapolis, Indiana
  - Phenomix Investigational Site 136, Brockton, Massachusetts
  - Phenomix Investigational Site 125, Kalamazoo, Michigan
  - Phenomix Investigational Site 138, Biloxi, Mississippi
  - Phenomix Investigational Site 122, Las Vegas, Nevada
  - Phenomix Investigational Site 140, Las Vegas, Nevada
  - Phenomix Investigational Site 131, Brick, New Jersey
  - Phenomix Investigational Site 110, Trenton, New Jersey
  - Phenomix Investigational Site 116, Albuquerque, New Mexico
  - Phenomix Investigational Site 107, Winston-Salem, North Carolina
  - Phenomix Investigational Site 130, Cincinnati, Ohio
  - Phenomix Investigational Site 118, Cuyahoga Falls, Ohio
  - Phenomix Investigational Site 112, Greenville, South Carolina
  - Phenomix Investigational Site 102, Dallas, Texas
  - Phenomix Investigational Site 139, Dallas, Texas
  - Phenomix Investigational Site 126, El Paso, Texas
  - Phenomix Investigational Site 104, San Antonio, Texas
  - Phenomix Investigational Site 100, Kenosha, Wisconsin
- Argentina (12):
  - Phenomix Investigational Site 401, Buenos Aires
  - Phenomix Investigational Site 402, Buenos Aires
  - Phenomix Investigational Site 404, Buenos Aires
  - Phenomix Investigational Site 405, Buenos Aires
  - Phenomix Investigational Site 406, Buenos Aires
  - Phenomix Investigational Site 407, Buenos Aires
  - Phenomix Investigational Site 408, Buenos Aires
  - Phenomix Investigational Site 409, Buenos Aires
  - Phenomix Investigational Site 411, Buenos Aires
  - Phenomix Investigational Site 403, Corrientes
  - Phenomix Investigational Site 410, Mendoza
  - Phenomix Investigational Site 400, Rosario
- Chile (5):
  - Phenomix Investigational Site 502, Santiago
  - Phenomix Investigational Site 504, Santiago
  - Phenomix Investigational Site 505, Santiago
  - Phenomix Investigational Site 500, Temuco
  - Phenomix Investigational Site 501, Temuco
- Czechia (9):
  - Phenomix Investigational Site 209, Chodov
  - Phenomix Investigational Site 205, Havířov-Město
  - Phenomix Investigational Site 204, Liberec
  - Phenomix Investigational Site 202, Olomouc
  - Phenomix Investigational Site 206, Ostrava-Kunčice
  - Phenomix Investigational Site 208, Prague
  - Phenomix Investigational Site 203, Prostějov
  - Phenomix Investigational Site 207, Uničov
  - Phenomix Investigational Site 201, Valašské Klobouky
- India (12):
  - Phenomix Investigational Site 703, Hyderabad, Andhara Pradesh
  - Phenomix Investigational Site 704, Visakhapatanam, Andhra Pradesh
  - Phenomix Investigational Site 709, Gopālapuram, Chennai
  - Phenomix Investigational Site 707, Shāstrinagar, Jaipur
  - Phenomix Investigational Site 701, Bangalore, Karnataka
  - Phenomix Investigational Site 702, Bangalore, Karnataka
  - Phenomix Investigational Site 705, Trivandrum, Kerala
  - Phenomix Investigational Site 706, Indore, Madhya Pradesh
  - Phenomix Investigational Site 711, Mumbai, Maharashtra
  - Phenomix Investigational Site 700, Nashik, Maharashtra
  - Phenomix Investigational Site 710, Navi Mumbai, Maharashtra
  - Phenomix Investigational Site 708, Chennai
- Peru (11):
  - Phenomix Investigational Site 607, Arequipa
  - Phenomix Investigational Site 601, Ica
  - Phenomix Investigational Site 600, Lima
  - Phenomix Investigational Site 603, Lima
  - Phenomix Investigational Site 604, Lima
  - Phenomix Investigational Site 608, Lima
  - Phenomix Investigational Site 610, Lima
  - Phenomix Investigational Site 605, Lima Cercado
  - Phenomix Investigational Site 606, Piura
  - Phenomix Investigational Site 602, Trujillo
  - Phenomix Investigational Site 609, Wanchaq Cusco
- Poland (14):
  - Phenomix Investigational Site 300, Gdansk
  - Phenomix Investigational Site 301, Gdansk
  - Phenomix Investigational Site 303, Katowice
  - Phenomix Investigational Site 312, Katowice
  - Phenomix Investigational Site 309, Krakow
  - Phenomix Investigational Site 313, Krakow
  - Phenomix Investigational Site 308, Lublin
  - Phenomix Investigational Site 310, Poznan
  - Phenomix Investigational Site 306, Puławy
  - Phenomix Investigational Site 304, Szczecin
  - Phenomix Investigational Site 305, Warsaw
  - Phenomix Investigational Site 307, Warsaw
  - Phenomix Investigational Site 311, Warsaw
  - Phenomix Investigational Site 302, Wroclaw